CLINICAL TRIAL: NCT02345018
Title: Registry of the Treatment of Primary Insufficiency of the Great Saphenous Vein With a Diameter >/= 12 mm, Antero-lateral Branches, or Great Saphenous Vein Insufficiency Below the Knee With Mechano-chemical Endovenous Ablation (MOCA)
Brief Title: Primary Insufficiency of the GSV With a Diameter >/= 12 mm, Antero-lateral Branches, or Below the Knee
Acronym: MOCA-XL
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, Vascular surgeon, Rijnstate Hospital
Other Study IDs: 1079-101114
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Varicose Veins; Dilated Veins
Keywords: Mechano-chemical ablation; Treatment large varicose veins; Below-knee and branches; Endovenous
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- GSV with diameters >/= 12 mm: 30 patients with primary insufficiency of the GSV with diameters >/= 12 mm, treated with mechano-chemical ablation (MOCA)
  Interventions: Procedure: Mechano-chemical ablation
- Antero-lateral branches: 30 patients with insufficient antero-lateral branches, treated with mechano-chemical ablation (MOCA)
  Interventions: Procedure: Mechano-chemical ablation
- GSV below-knee: 30 patients with below-knee GSV insufficiency, treated with mechano-chemical ablation (MOCA)
  Interventions: Procedure: Mechano-chemical ablation

INTERVENTIONS:
Procedure: Mechano-chemical ablation — Treatment with mechano-chemical ablation
  Other Names: MOCA

SUMMARY:
The goal of this registry study is to provide insight in the safety and efficacy of treatment with MOCA for primary insufficiency of the GSV with a diameter >/=12mm, insufficient antero-lateral branches and insufficiency of the GSV below the knee.

DETAILED DESCRIPTION:
Varicose veins are a common problem in the World. From epidemiological studies we know that a quarter of the adult population suffers from some sort of varicose veins. Women suffer two to three times more often from varicose veins than men. The occurrence of varicose veins increase with increasing age and is one of the top ten complaints for which patients visit their general practitioner. De main risk factors for developing varicose veins are enduring standing or sitting, pregnancy, female gender and age. Symptoms are divers and vary from cosmetic complaints to difficult to treat venous ulcers.

Last few years endovenous techniques have been developed for the primary treatment of insufficient varicose veins. Radiofrequent ablation (RFA)is, besides endovenous laser ablation (EVLA), an accepted technique and is frequently applied in clinical practice. This technique, that uses heat, has the important advantage that the treatment can be performed using a slight local anaesthesia. Besides that, RFA causes less hematoma, pain, a superior cosmetic and patient are able to restart daily activities sooner than compared to the classical surgical treatment. Because RFA using heat technology, damage can occur in the surrounding tissues. That is the reason for using tumescent anaesthesia, for which multiple injections are needed. A column of liquid is placed surrounding the vein. Many patients experience this column as inconvenient and despite this form of anaesthesia part of the treated patient population experiences pain after the treatment that can last up to weeks.

A newer endovenous technique is mechano-chemical ablation (MOCA) has been developed, using the ClariVein system. This technique uses intentional mechanical damage to the endothelium of the vene by means of a rotating catheter. At the same time a sclerosans is injected, and as a result the vene occludes. So this technique does not use heat technology. Tumescent anaesthesia is therefore not needed and complications related to techniques using heat (RFA and EVLA) such as burning, pain, hematoma, indurations, and paresthesia could be reduced or even be prevented.

MOCA proved to be a safe and effective alternative treatment for both insufficient great saphenous veins (GSV) and small saphenous veins (SSV). Especially for the treatment of the below-knee GSV and the treatment of superficial branches (such as the antero-lateral branches), there is a risk for damaging nerves that are in the close proximity of these veins.

In a series of 50 patients treated with EVLA for insufficient GSV above the knee, a technical success of 100% was reported after a median follow-up of 7 months, but this was accompanied by nerve damage in 8%. A recent study evaluating MOCA for the treatment of SSV reported an anatomical success of 96% without any nerve damage or other major complications. Therefore, MOCA could be an alternative for the treatment of various insufficient varicose vein segments without causing nerve damage.

The choice of treatment for patients with both above and below knee GSV insufficiency is nowadays only endovenous ablation of the above-knee segment. However, Theivacumar and co-workers recently showed that in these patients there is a significant residual reflux in approximately 41% of treated legs. These patients clearly showed less clinical improvement and approximately 90% of these patients needed additional treatment.

Up to now it is unknown whether treatment with MOCA can yield comparable results when used to treat insufficient GSV with diameters >= 12 mm, insufficient antero-lateral branches and insufficient GSV below the knee. The goal of this registry study is to provide insight in the safety and efficacy of treatment of the above described insufficient varicose vein segments.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic varicose veins, C2-C5
2. Ultrasound criteria:

   1. Diameter supragenual great saphenous vein (GSV) >/= 12 mm , not tortuous; or
   2. Insufficient antero-lateral branch; or
   3. Insufficient below knee GSV
3. Signed informed consent
4. Patient consents to follow-up
5. Age > 18 year en < 80 year

Exclusion Criteria:

1. Patient is not capable to provide informed consent
2. Pregnancy and lactation
3. C6 varicose veins
4. Previous surgery or endovenous ablation at to treated segment
5. Deep venous vein thrombosis in medical history
6. Oral anti-coagulant therapy
7. Contra-indications or allergy for sclerosant
8. Immobilisation
9. Coagulant disorders or increased risk for thrombo-embolic complications: known coagulant disorders such as hemophilia A, hemophilia B, Von Willebrand disease, Glanzmann disease, factor VII-deficiency, idiopathic thrombo-cytopenic purpura, factor V Leiden disease and deep venous thrombosis or lung emboli in medical history
10. Fontaine III of IV peripheral arterial disease
11. Severe kidney disease: known GFR < 30 ml/min
12. Liver diseases accompanied by changes in coagulation of the blood, anamnestic indications for tendency towards haemorrhage , such as epistaxis and spontaneous hematoma, known liver cirrhosis

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary insufficiency of the GSV with diameters >/=12 m m, insufficient antero-lateral branches or below-knee GSV insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-06; Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Anatomical success | 4 weeks + 1 year
  Occlusion rate, evaluated using ultrasound scan
Clinical success | 4 weeks + 1 year
  CEAP, VCSS
Peroperative pain | Peroperative
  VAS-score
Postoperative pain during 2 weeks post-treatment | During 2 weeks post-treatment
  VAS-score, used pain medication

SECONDARY OUTCOMES:
Postoperative complications | 4 weeks + 1 year
  Postoperative complications
Disease specific and general health status | 4 weeks + 1 year
  AVVQ, SF-36
Time to return to normal daily activities and work | Post-treatment
  Time to return to normal daily activities and work
Duration of the intervention using MOCA | Peroperative
  Duration of the intervention using MOCA

CONTACTS AND LOCATIONS:
Overall Officials: Michel Reijnen, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Background] Rasmussen LH, Bjoern L, Lawaetz M, Blemings A, Lawaetz B, Eklof B. Randomized trial comparing endovenous laser ablation of the great saphenous vein with high ligation and stripping in patients with varicose veins: short-term results. J Vasc Surg. 2007 Aug;46(2):308-15. doi: 10.1016/j.jvs.2007.03.053. Epub 2007 Jun 27. PMID 17600655
- [Background] Helmy ElKaffas K, ElKashef O, ElBaz W. Great saphenous vein radiofrequency ablation versus standard stripping in the management of primary varicose veins-a randomized clinical trial. Angiology. 2011 Jan;62(1):49-54. doi: 10.1177/0003319710380680. Epub 2010 Aug 18. PMID 20724299
- [Background] Subramonia S, Lees T. Randomized clinical trial of radiofrequency ablation or conventional high ligation and stripping for great saphenous varicose veins. Br J Surg. 2010 Mar;97(3):328-36. doi: 10.1002/bjs.6867. PMID 20035541
- [Background] van Eekeren RR, Boersma D, Elias S, Holewijn S, Werson DA, de Vries JP, Reijnen MM. Endovenous mechanochemical ablation of great saphenous vein incompetence using the ClariVein device: a safety study. J Endovasc Ther. 2011 Jun;18(3):328-34. doi: 10.1583/11-3394.1. PMID 21679070
- [Background] Boersma D, van Eekeren RR, Werson DA, van der Waal RI, Reijnen MM, de Vries JP. Mechanochemical endovenous ablation of small saphenous vein insufficiency using the ClariVein((R)) device: one-year results of a prospective series. Eur J Vasc Endovasc Surg. 2013 Mar;45(3):299-303. doi: 10.1016/j.ejvs.2012.12.004. Epub 2013 Jan 9. PMID 23312507
- [Background] Bishawi M, Bernstein R, Boter M, Draughn D, Gould CF, Hamilton C, Koziarski J. Mechanochemical ablation in patients with chronic venous disease: a prospective multicenter report. Phlebology. 2014 Jul;29(6):397-400. doi: 10.1177/0268355513495830. Epub 2013 Jul 2. PMID 23820117
- [Background] van Eekeren RR, Boersma D, Konijn V, de Vries JP, Reijnen MM. Postoperative pain and early quality of life after radiofrequency ablation and mechanochemical endovenous ablation of incompetent great saphenous veins. J Vasc Surg. 2013 Feb;57(2):445-50. doi: 10.1016/j.jvs.2012.07.049. Epub 2012 Nov 8. PMID 23141679
- [Background] Timperman PE. Endovenous laser treatment of incompetent below-knee great saphenous veins. J Vasc Interv Radiol. 2007 Dec;18(12):1495-9. doi: 10.1016/j.jvir.2007.07.029. PMID 18057283
- [Background] Theivacumar NS, Dellagrammaticas D, Mavor AI, Gough MJ. Endovenous laser ablation: does standard above-knee great saphenous vein ablation provide optimum results in patients with both above- and below-knee reflux? A randomized controlled trial. J Vasc Surg. 2008 Jul;48(1):173-8. doi: 10.1016/j.jvs.2008.01.062. Epub 2008 Apr 28. PMID 18440756